CLINICAL TRIAL: NCT02269254
Title: Migration and Kinematics of the New Persona PS Versus the Proven NexGen LPS Knee - a Randomized Controlled Trial Using Radiostereometric Analysis and Fluoroscopy
Brief Title: Persona Versus NexGen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, R.G.H.H. Nelissen, Prof. PhD MD Head of the Department of Orthopaedics, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P13.277
Record Dates: First submitted 2014-09-23; First posted 2014-10-21 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Comparative Study; Knee Prosthesis; Prosthesis Design; Treatment Outcome; Follow-Up Studies; Arthroplasty, Replacement, Knee/methods
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Persona PS (Experimental): Total Knee Replacement with Persona PS Knee Prosthesis by Zimmer
  Interventions: Device: Persona PS Knee Prosthesis by Zimmer
- NexGen PS (Active Comparator): Total Knee Replacement with NexGen PS Knee Prosthesis by Zimmer
  Interventions: Device: NexGen PS Knee Prosthesis by Zimmer

INTERVENTIONS:
Device: Persona PS Knee Prosthesis by Zimmer — Total Knee Replacement with Persona PS Knee Prosthesis by Zimmer
  Arms: Persona PS
Device: NexGen PS Knee Prosthesis by Zimmer — Total Knee Replacement with NexGen PS Knee Prosthesis by Zimmer
  Arms: NexGen PS

SUMMARY:
The NexGen TKR (Zimmer, Warsaw, Indiana, USA) is a proven TKR design that has reported excellent medium and long-term results in clinical studies and in implant registries all around the world. As a follow-up of the NexGen TKR, an improved design has recently been introduced by Zimmer: The Persona TKR (Zimmer, Warsaw, Indiana, USA) has been used successfully in about 20.000 patients, but results from independent clinical studies have not been reported yet.

The objective of this study is to accurately assess and compare migration, kinematics, prosthesis placement and patient reported outcomes of two TKR prostheses: the fixed bearing, cemented NexGen LPS, a proven design with an excellent clinical track record, and the fixed bearing, cemented Persona PS, a new design without clinical data (both designs by Zimmer, Warsaw, Indiana, USA). The primary objective is to assess and compare migration of the two TKR prostheses (Femoral and Tibial component). The secondary objective is to assess and compare clinical data, kinematics, prosthesis placement and patient reported outcome measures.

This study is designed as a single-blind randomized trial between the Persona PS total knee prosthesis and the well-established NexGen total knee prosthesis.

Different sample sizes are used for the different parts of this study:

* 30 Patients with NexGen LPS prosthesis and 30 patients with Persona PS prosthesis for RSA
* 15 Patients with NexGen LPS prosthesis and 15 patients with Persona PS prosthesis for Fluo

The study population will consist of patients with symptomatic osteoarthritis of the knee scheduled for TKR surgery at the Department of Orthopaedics, Leiden University Medical Center. Annually 40 TKA procedures are performed in our department, of which about 70% is Osteo Arthritis (OA) and 30% Reumatoid Arthritis (RA). We anticipate that inclusion can be accomplished within a 2 year period.

Main study parameters/endpoints are:

* Migration, measured by means of RSA.
* Prosthesis placement and bone resection measured by means of CT and caliper measurements of the resected bone parts.
* In vivo kinematics by means of fluoroscopy.
* Patient Reported Outcome Measures by means of questionaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with osteoarthritis or rheumatoid arthritis and requiring primary knee arthroplasty
* Patient has been classified ASA 1 or 2 (for the kinematic analysis) (Meyer Saklad, 1941). As for the RSA study all consecutive patients ("usual care") are included to prevent selection bias in the migration analysis. Stratification is performed per diagnosis group (OA/RA).

Exclusion Criteria:

* The patient is unable or unwilling to sign the Informed Consent specific to this study
* Insufficient Dutch or English language skills
* Patients indicated for revision arthroplasty
* Patient is (or might be) pregnant
* When there are less than five tibia-bone markers and less than five femur-bone markers visible in the baseline RSA photograph and it will not improve by placing the patient in another position, the patient will be excluded from the study (secondary exclusion criteria). In case only one of the bones has insufficient markers, the patient will be followed for the other bone.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Migration, measured by means of RSA. | 2 Years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA).

SECONDARY OUTCOMES:
Knee Prosthesis motion by means of Fluoroscopy. | 1 Year
  Motion of the knee prosthesis during a step-up movement, measured by means of Fluoroscopic Motion Analysis.
EQ-5D | 2 Years
  General Health: EuroQol 5 Dimensional (EQ-5D) Health Questionnaire measured using patient questionnaire
KOOS | 2 Years
  Knee Function: Knee injury and Osteoarthritis Outcome Score (KOOS) measured using patient questionnaire
VAS pain | 2 Years
  Pain score after activity and during rest; (Likert scale 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Rob GHH Nelissen, Prof. PhD, MD, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center; Edward R Valstar, Prof. PhD. MSc, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands